CLINICAL TRIAL: NCT04317703
Title: A Randomized, Open-label, Single-dose, Two-way Crossover Bioequivalence Study of Fixed Dose Combination Zemimet® SR Tab. 50/1000 mg (Gemigliptin/Metformin Hydrochloride Sustained Release 50/1000 mg) and Coadministration of Zemiglo Tablet 50 mg (Gemigliptin 50 mg) and Glucophage® XR 1000 mg (Metformin Hydrochloride Prolonged Release 1000 mg) Under Fasting Conditions in Healthy Volunteers
Brief Title: Bioequivalence Study for Fixed Dose Combination Zemimet® SR Tab. 50/1000 and Coadministration of Gemigliptin 50 mg and Metformin 1000 mg.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LG-DMCL009
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; LC15-0444

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test: Gemigliptin/Metformin (Experimental): Fixed Dose Combination Zemimet® SR Tab. 50/1000 mg (Gemigliptin/Metformin Hydrochloride Sustained Release 50/1000 mg)
  Interventions: Drug: Gemigliptin tartrate sesquihydrate and metformin
- Reference: Gemigliptin and Metformin (Active Comparator): Coadministration of Zemiglo Tablet 50 mg (Gemigliptin 50 mg) and Glucophage XR 1000 mg (Metformin Hydrochloride Prolonged Release 1000 mg)
  Interventions: Drug: gemigliptin 50 mg and metformin hydrochloride 1000 mg prolonged release

INTERVENTIONS:
Drug: Gemigliptin tartrate sesquihydrate and metformin — Each tablet contains gemigliptin tartrate sesquihydrate 68.9 mg (equivalent to gemigliptin pure free base 50 mg) and metformin hydrochloride 1000.0 mg.
  Other Names: Zemimet® SR Tab. 50/1000 mg
  Arms: Test: Gemigliptin/Metformin
Drug: gemigliptin 50 mg and metformin hydrochloride 1000 mg prolonged release — Zemiglo Tablet 50 mg: Each tablet contains gemigliptin tartrate sesquihydrate, equivalent to 50 mg gemigliptin.
  Glucophage XR 1000 mg: Each tablet contains metformin hydrochloride 1000 mg (equivalent to 780 mg of metformin base).
  Other Names: Zemiglo Tablet 50 mg and Glucophage XR 1000 mg
  Arms: Reference: Gemigliptin and Metformin

SUMMARY:
To determine and compare the rate and extent of absorption of gemigliptin/metformin hydrochloride sustained release 50/1000 mg FDC tablet (Zemimet® SR Tab. 50/1000 mg) and coadministration of corresponding dose of gemigliptin 50 mg (Zemiglo Tablet 50 mg) and metformin hydrochloride 1000 mg prolonged release (Glucophage XR 1000 mg) as individual tablet in healthy subjects under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18.0 to 30.0 kg/m2.
* Normal laboratory values, including vital signs and physical examination, for all parameters in clinical laboratory tests at screening.
* Non-pregnant woman (negative pregnancy test) and not currently breast feeding
* Female subjects abstain from either hormonal methods of contraception
* Male subjects who are willing or able to use effective contraceptive
* Have voluntarily given written informed consent (signed and dated) by the subject prior to participating in this study.

Exclusion Criteria:

* History serious hypersensitivity reactions
* History or evidence of clinically significant diseases or any significant ongoing chronic medical illness
* History or evidence of family diabetes
* History or evidence of type 1 diabetes mellitus, diabetic ketoacidosis, diabetic pre-coma
* History or evidence of shock or severe dehydrate or severe infection
* History or evidence of preceding diarrhea or vomiting within 24 hours prior to admission in each period
* History or evidence of drug addict or investigation with urine sample shows a positive test for drug of abuse
* History of problems with swallowing tablet or capsule
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* Any condition possibly affecting drug absorption
* Have renal creatinine clearance (Clcr) < 45 mL/min based on serum creatinine results at the screening laboratory test
* 12-lead ECG demonstrating QTc >450 msec, a QRS interval >120 msec or with an abnormality considered clinically significant at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2020-09-05 (Actual); Study Completion 2020-09-05 (Actual)

PRIMARY OUTCOMES:
bioequivalence study | Blood samples (10 mL each) will be collected at time 0.00 (pre-dose; 2x10 mL in duplicate tubes) and at 0.50, 1.00, 1.50, 2.00, 3.00, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 14.00, 24.00, 32.00 and 48.00 hours post-dose
  To determine and compare the rate and extent of absorption of gemigliptin/metformin hydrochloride sustained release 50/1000 mg FDC tablet (Zemimet® SR Tab. 50/1000 mg) and coadministration of corresponding dose of gemigliptin 50 mg (Zemiglo Tablet 50 mg) and metformin hydrochloride 1000 mg prolonged release (Glucophage XR 1000 mg) as individual tablet in healthy subjects under fasting conditions

CONTACTS AND LOCATIONS:
Overall Officials: Porrani Puranajoti, Ph.D, Principal Investigator — International Bio Service Co., Ltd.
Locations (1):
- International Bio Service Co., Ltd., Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: No